CLINICAL TRIAL: NCT01979068
Title: Vascular Inflammation Stratified by Body Size Phenotype
Status: Completed | Type: Observational
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, K. M. Choi, Professor, Korea University
Other Study IDs: PET_MONW
Record Dates: First submitted 2013-10-28; First posted 2013-11-08 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Atherosclerosis; Obesity; Metabolic Syndrome
MeSH Terms: conditions — Atherosclerosis; Obesity; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
* Vascular Inflammation is a key factor in both the pathogenesis and outcome of atherosclerosis. 18FDG-PET is a promising novel tool for identifying and quantifying vascular inflammation within atherosclerotic plaque
* Recently, unique subsets of obese individuals, such as metabolically obese but normal weight (MONW) and metabolically healthy obese (MHO), have been getting an attention
* Therefore, the purpose of this study is to examine the relationship of vascular inflammation,measured by FDG-PET, with various body sized phenotypes

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients for visiting routine medical check in our clinic

Exclusion Criteria:

* history of CVD (myocardial infarction, unstable angina, stroke, or cardiovascular revascularization)
* stage 2 hypertension (resting blood pressure, ≥160/100 mmHg)
* history of inflammatory conditions that affect the study results
* taking medications that might affect inflammatory status, including steroid and non-steroidal anti-inflammatory drug within 6 months
* or malignancy or severe renal or hepatic disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers who underwent a medical health check in the health promotion center in Korea University Guro Hospital
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2008-03; Primary Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
max TBR values stratified by the four body size phenotypes | 12 weeks

SECONDARY OUTCOMES:
Framingham risk scores according to the four body size phenotypes | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Yoo HJ, Kim S, Hwang SY, Hong HC, Choi HY, Seo JA, Kim SG, Kim NH, Choi DS, Baik SH, Choi KM. Vascular inflammation in metabolically abnormal but normal-weight and metabolically healthy obese individuals analyzed with (1)(8)F-fluorodeoxyglucose positron emission tomography. Am J Cardiol. 2015 Feb 15;115(4):523-8. doi: 10.1016/j.amjcard.2014.11.036. Epub 2014 Nov 29. PMID 25529544